CLINICAL TRIAL: NCT05502185
Title: Targeting Staphylococci Adhesion and Colonization on the Surface of Corneocytes in Atopic Dermatitis
Brief Title: Targeting Staphylococci in Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Other Study IDs: ACR_TCDUB_22-11995
Record Dates: First submitted 2022-07-12; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Bacterial adhesion
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — corneocytes (stratum corneum upper layer of the dead skin part without nucleus and DNA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: no intervention
- Atopic Dermatitis patients: no intervention

SUMMARY:
The aim of the study is to deliver a better understanding of the molecular mechanisms used by S. epidermidis strains in their adhesion and colonization on the stratum corneum across a broad spectrum of atopic dermatitis in mild to moderate conditions in adult patients.

DETAILED DESCRIPTION:
Recent studies have shown that while in severe cases of AD the density of S. aureus is increased in lesions, the skin of adult patients with low to mild AD were overpopulated with S. epidermidis and not S. aureus.

the aim is to characterize the S. epidermidis colonization and adhesion, with the Analyzis of skin and microbiota samples to identify and characterize S. epidermidis strains involved in corneocytes adhesion.

ELIGIBILITY:
Inclusion Criteria:

* • Male/Female subject from 18 years old or above.

  * Subject willing and able to fulfil the study requirements and schedule
  * Subject informed about the study objectives and procedures, and able to understand them
  * Subject who has given written informed consent
  * Subject with I, II, III or IV skin phototype
  * Specific criteria:

For AD patients:

* Subject diagnosed with AD (via UK working party criteria) with a mild-to-moderate severity defined as EASI<32 and vIGA between 2 and 3
* Subject with at least one AD lesion covering at least 4 cm²

For healthy volunteers:

• Subject matching the demographic characteristics of a patient included in the AD group: same sex, same phototype, same age (± 5 years)

Exclusion Criteria:

* Subject with a body mass index (BMI) higher than 40
* Presenting another dermatological condition that could interfere with the clinical evaluation
* Presenting any concomitant medical condition that may interfere with the study conduct in the opinion of the investigator
* Topical or systemic treatment that could interfere with the study treatment/assessments (topical benzoyl peroxide, salicylic acid and other anti-acne or antiseborrheic products, antibiotics, corticosteroids, retinoids, differin gel, retin-A, anti-inflammatory drugs, within the 4 weeks prior to the participation in the study.
* Any physical treatment including laser or phototherapy (PUVA, IPL, PDT), topical fillers such as Botox on the investigational sites in the last 6 months and during the study
* Subject treated with systemic non-steroidal anti-inflammatory drugs (≥3 days) within 1 week before the inclusion visit or intending to be treated with it during the study.
* Subject treated with biological immunosuppressive drugs within 12 weeks prior to the inclusion visit or intending to be treated with it during the study.
* Subject treated with non-biological immunosuppressive drugs within 4 weeks prior to the inclusion visit or intending to be treated with it during the study.
* Subject treated with systemic corticoids within 1 week prior to the inclusion visit or planed during the study.
* Subject treated with systemic antibiotics within 2 weeks prior to the inclusion visit or planned during the study.
* Subject having applied topical corticosteroids and topical calcineurin inhibitors on the investigational areas within 1 week prior to the inclusion visit.
* Subject having applied topical immunomodulators, non-steroidal anti-inflammatory, antihistamines on investigational area within 1 week prior to the inclusion visit.
* Subject having applied topical antibiotics or disinfectants on investigational area within 2 weeks prior to the inclusion visit.
* Subject having applied any other topical and/or care product within 12 hours of the visit.
* Subject having applied water or care product (except hands cleaning) within 12 hours prior to the inclusion visit.
* Subject having significant dermatological condition or sign (e.g disease, scare, abundant hairiness, tanning mark…) that according to the investigator's judgment, could limit the observations or/and interfere with the interpretations.
* Subject having performed phototherapy within 8 weeks prior to the inclusion visit or intending to perform phototherapy during the study.
* Subject having performed another physical treatment (e.g radiotherapy…) on the investigational areas within 6 months prior to the inclusion visit or intending to perform it during the study.
* Subject having exposed their skin to natural or artificial UV within 2 weeks prior to the inclusion visit
* Subject under legal guardianship or incapacitation.
* Subject who declares to be deprived of freedom by administrative or legal decision
* Subject linguistically or psychologically unable of signing informed consent form and unable to comply with the protocol requirements according to the investigator's judgment.
* Subject who cannot be contacted by telephone in case of emergency.
* Subject having participated within the 30 days before inclusion or currently participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 participants (30 healthy volunteers and 30 AD patients)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Identification of S. epidermidis adhesins | 1 week
  Identification of S. epidermidis adhesins involved in corneocytes adhesion, in mild-to moderate AD conditions

SECONDARY OUTCOMES:
characterization of corneocytes | 1 week
  characterization of corneocytes morphology from clinical sourcing of lesional and non lesional zones of AD subjects, mild-to-moderate and healthy volunteers, and characterization of the interaction between S. epidermidis adhesins and AD corneocytes

CONTACTS AND LOCATIONS:
Overall Officials: Alan IRVINE, MD, Principal Investigator — Clinical Research Facility in Trinity College of Dublin/St. James Hospital

IPD SHARING:
Plan to Share IPD: No